CLINICAL TRIAL: NCT01026467
Title: A Phase II Study of Fraility Index and Geriatric Assessment as Predictors of Toxicity to Front-Line Chemotherapy in Patients With Stage IV Non-Small Cell Lung Cancer
Brief Title: Frailty Index and Geriatric Assessment in Predicting Toxicity to Front-Line Chemotherapy in Treating Patients With Stage IV Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00011804; NCI-2009-01451 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 98709 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Carboplatin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Supportive Care (frailty index, geriatric assessment, chemo): Patients complete a frailty index and geriatric assessment prior to beginning chemotherapy. Patients receive standard-of-care chemotherapy comprising carboplatin IV and paclitaxel IV on day 1. Treatment repeats every 21 days for up to 2 courses
  Interventions: Drug: cisplatin; Drug: carboplatin; Other: questionnaire administration

INTERVENTIONS:
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Other: questionnaire administration

SUMMARY:
This phase II trial is studying how well a frailty index and geriatric assessment works in predicting toxicity to front-line chemotherapy in treating patients with stage IV non-small cell lung cancer. A frailty index and geriatric assessment prior to treatment may help identify a better treatment regimen

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the correlation of the data from the frailty index and geriatric assessment tool with the level of toxicity encountered in the first two cycles of therapy.

OUTLINE:

Patients complete a frailty index and geriatric assessment prior to beginning chemotherapy. Patients receive standard-of-care chemotherapy comprising carboplatin intravenously (IV) and paclitaxel IV on day 1. Treatment repeats every 21 days for up to 2 courses.

ELIGIBILITY:
Inclusion Criteria:

Pathological documentation of non-small cell lung cancer Stage IV disease Prior adjuvant chemotherapy for the earlier stages of non-small cell lung cancer is allowed Patients with brain metastases are allowed on protocol only if they have received brain irradiation and are neurologically stable Patients with other malignancies are allowed on protocol unless they are receiving active treatment (surgery, radiation, chemotherapy or immunotherapy) for the other malignancy Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

Prior palliative chemotherapy Pregnant and/or lactating women Prior radiation therapy other than brain irradiation for brain metastases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Stage IV Non-Small Cell Lung Cancer
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Use of the Frailty Index and/or the geriatric assessment in prediction of toxicity | Prior to chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Klepin, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Syracuse VA Medical Center, Syracuse, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina